CLINICAL TRIAL: NCT01008449
Title: Surgical Staples vs. Absorbable Subcuticular Suture for Wound Closure of Cesarean Deliveries
Brief Title: Staples Versus Suture for Cesarean Wound Closure
Acronym: SVS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New studies were reporting that sutures are beneficial, hindering the possibility of enrollment.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Alan Tita, Physician, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X090531008
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Wound
Keywords: Staples; Sutures; Cesarean Delivery; Wound; Skin Closure; Wound infection; Wound disruption
MeSH Terms: conditions — Wounds and Injuries; Wound Infection | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Absorbable Subcuticular Surgical Suture (Active Comparator): Patients in this arm will receive absorbable subcuticular suture for wound closure of cesarean deliveries.
  Interventions: Device: Absorbable Surgical Suture
- Surgical staples (Active Comparator): Patients in this arm will receive surgical staples for wound closure.
  Interventions: Device: Surgical staples

INTERVENTIONS:
Device: Surgical staples — Surgical staples will be used once for wound closure.
  Other Names: Proximate Plus MD 35 W, Ethicon Endo-surgery
  Arms: Surgical staples
Device: Absorbable Surgical Suture — Absorbable surgical suture will be used for subcuticular closure at the time of wound closure for cesarean delivery.
  Other Names: 4-0 Monocryl, Ethicon
  Arms: Absorbable Subcuticular Surgical Suture

SUMMARY:
The objective of this randomized controlled trial is to compare wound morbidity (including disruption and infection) in surgical staples versus absorbable subcuticular suture for wound closure in cesarean deliveries.

DETAILED DESCRIPTION:
Cesarean delivery (CD) is a common surgical procedure with over 1 million performed annually in the United States. The rate of CD is steadily increasing. In 2006, an estimated 31.1% of U.S. births were by CD. Approximately two thirds of these are primary procedures and 90% of CD will later undergo a repeat cesarean delivery. The rise in CD has been attributed to changes in physician and patient expectations, attitudes about risk, and changes in clinical practice. These include decreased vaginal birth after cesarean delivery (VBAC), breech vaginal deliveries, and operative vaginal deliveries as well as an increase in maternal request, failed induction of labor, and elective repeat CD. The CD rate is expected to rise as high as 40-50% in the next decade if the increasing trend continues unabated.

Despite the large number of CD performed, there is no agreed standard for skin closure. The most commonly used materials are surgical staples and absorbable subcuticular suture. Staples have a clear benefit in decreasing operating time. In theory, staples also have a decreased chance of bacterial migration into the wound, decreased tension at the incision edges, and less damage to capillaries in the subcuticular layer of skin than absorbable subcuticular suture. However, some argue that staples are more painful and have a worse cosmetic appearance. This is especially the case for staples that remain in place longer than recommended and leave "track marks." Staples are also less visually appealing to patients.

The Cochrane Collaboration identified one randomized controlled trial (RCT) that addressed skin closure for CD (Alderice, 2003). This study included 66 women and compared absorbable subcuticular suture versus surgical staples for skin closure of CD. Surgical staples had shorter operating time but absorbable subcuticular suture had decreased post-operative pain and better cosmesis at the 6 week post-operative visit (Frishman, 1997). Rousseau, J. presented opposing findings in her RCT "A Randomized Study Comparing Subcuticular Sutures Versus Staples for Skin Closure at Cesarean Sections". In this study, staples had better cosmesis, decreased pain at the post-operative visit, and shorter operating time (Rousseau, 2009). Neither study assessed wound disruption or infection directly. With such widely varying findings and lack of data there is a need to identify the cesarean section skin closure which provides the best outcomes for the most common major surgical procedure in women.

We have undertaken a RCT to compare surgical staples vs. absorbable subcuticular suture for the closure of the skin in cesarean sections. Our primary outcome is a composite wound morbidity outcome (including wound disruption or infection). Assuming a baseline wound morbidity of 8%, Power of 80%, and a decrease of wound morbidity to 4%, a sample size of 1,204 will be required. Our secondary outcomes will include cosmesis, post-operative pain, health service use/cost, procedure time, and patient satisfaction.

The study was terminated after recruitment of approximately 400 subjects after administrative review (see publication: Figueroa et al. Obstet Gynecol. 2013 Jan;121(1):33-8.)

ELIGIBILITY:
Inclusion Criteria:

* cesarean delivery

Exclusion Criteria:

* chronic use of immunosuppressive agents ( e.g.po steroids > 2 weeks)
* significant immune compromising disease (e.g. AIDS, CD4<200)
* contraindication to standard post operative pain management (acetaminophen, ibuprofen, oxycodone)
* refusal or inability to give consent

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2009-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Figueroa, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Hospital, Birmingham, Alabama, United States

REFERENCES:
- [Background] Rousseau JA, Girard K, Turcot-Lemay L, Thomas N. A randomized study comparing skin closure in cesarean sections: staples vs subcuticular sutures. Am J Obstet Gynecol. 2009 Mar;200(3):265.e1-4. doi: 10.1016/j.ajog.2009.01.019. PMID 19254586
- [Background] Frishman GN, Schwartz T, Hogan JW. Closure of Pfannenstiel skin incisions. Staples vs. subcuticular suture. J Reprod Med. 1997 Oct;42(10):627-30. PMID 9350017
- [Background] Alderdice F, McKenna D, Dornan J. Techniques and materials for skin closure in caesarean section. Cochrane Database Syst Rev. 2003;(2):CD003577. doi: 10.1002/14651858.CD003577. PMID 12804476
- [Derived] Figueroa D, Jauk VC, Szychowski JM, Garner R, Biggio JR, Andrews WW, Hauth J, Tita AT. Surgical staples compared with subcuticular suture for skin closure after cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2013 Jan;121(1):33-8. doi: 10.1097/aog.0b013e31827a072c. PMID 23262925
- See also: Link to study results on PubMed — http://www.ncbi.nlm.nih.gov/pubmed/23262925

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Absorbable Subcuticular Surgical Suture | Surgical Staples
Started | 200 | 198
Completed | 171 | 179
Not Completed | 29 | 19
Not completed — Lost to Follow-up | 29 | 19

BASELINE CHARACTERISTICS:
Population: subjects that that were lost to follow up were not included in the results
Groups:
- Total: Total of all reporting groups
Arm/Group | Absorbable Subcuticular Surgical Suture | Surgical Staples | Total
Number analyzed (Participants) | 171 | 179 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (5.9) | 26.7 (6.1) | 26.8 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 179 | 350
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 171 | 179 | 350

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With Composite Wound Morbidity.
Description: this outcome measure included a composite of either disruption and/ or infection of the wound at 4 - 6 weeks post partum. The number of subjects experiencing wound disruption and or wound infection at 4 - 6 weeks post delivery was assessed
Time Frame: 4-6 weeks post partum
Measure: Number; unit: percentage of subjects
Arm/Group | Absorbable Subcuticular Surgical Suture | Surgical Staples
Number analyzed (Participants) | 171 | 179
percentage of subjects | 5.9 | 14.5

2. Secondary Outcome: Composite Cosmesis Score (Stony Brook Scar Evaluation Score - SBSES) Core - SBSES))
Description: The SBSES assessed five scar components: width, height, color, suture marks and overall appearance. Each component was assigned a score of 0 or 1 with a total sum range of 0 (worst) to 5 (best).
Time Frame: at the end of follow up, 4 - 6 weeks post partum
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Absorbable Subcuticular Surgical Suture | Surgical Staples
Number analyzed (Participants) | 171 | 179
units on a scale | 4 [3 to 5] | 3 [3 to 4]

3. Secondary Outcome: Operative Procedure Time.
Description: time for procedure as measured in minutes
Time Frame: Intraoperative, at time of intervention.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Absorbable Subcuticular Surgical Suture | Surgical Staples
Number analyzed (Participants) | 171 | 179
minutes | 40 [28 to 55] | 37 [29 to 53]

4. Secondary Outcome: Post Operative Pain - 4 - 6 Weeks Post Delivery
Description: the visual analog pain scale was used. The range is 0 to 10 for reporting pain: 0 = no pain and 10 = unbearable distress
Time Frame: at end of follow-up, 4 - 6 weeks post partum
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Absorbable Subcuticular Surgical Suture | Surgical Staples
Number analyzed (Participants) | 171 | 179
units on a scale | 0 [0 to 2] | 0 [0 to 1]

5. Secondary Outcome: Post Operative Pain - 72 - 96 Hours Post Delivery
Description: as for outcome 4
Time Frame: 72 - 96 hours post delivery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Absorbable Subcuticular Surgical Suture | Surgical Staples
Number analyzed (Participants) | 171 | 179
units on a scale | 5 [4 to 7] | 5 [3 to 7]

6. Secondary Outcome: Subject Reported Satisfaction With Appearance of Scar
Description: Subject reported satisfaction of the scar appearance was assessed by using a scale of 1 - 5 with 1 being worst appearance and 5 being best appearance
Time Frame: 4 - 6 weeks post delivery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Absorbable Subcuticular Surgical Suture | Surgical Staples
Number analyzed (Participants) | 171 | 179
units on a scale | 4 [4 to 5] | 4 [4 to 5]

7. Secondary Outcome: Subject Satisfaction With Comfort With Scar
Description: Scar discomfort satisfaction was reported by subject perception using a scale of 1 - 5. A score of 1 would be the worst comfort and a score of 5 would be the best comfort
Time Frame: at end of follow-up, 4 - 6 weeks post partum
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Absorbable Subcuticular Surgical Suture | Surgical Staples
Number analyzed (Participants) | 171 | 179
units on a scale | 4 [4 to 5] | 4 [4 to 5]

8. Secondary Outcome: Subject Satisfaction With Location of Scar
Description: Satisfaction with location of scar was reported by subject using a scale of 1 - 5. A score of 1 would be the worst location of a scar and a score of 5 would be the best location of a scar
Time Frame: at end of follow-up, 4 - 6 weeks post partum
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Absorbable Subcuticular Surgical Suture | Surgical Staples
Number analyzed (Participants) | 171 | 179
units on a scale | 4 [4 to 5] | 4 [4 to 5]

ADVERSE EVENTS:
Arm/Group | Absorbable Subcuticular Surgical Suture | Surgical Staples
Serious Adverse Events (participants affected / at risk) | 0/171 | 0/179
Other Adverse Events (participants affected / at risk) | 12/171 | 28/179
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Absorbable Subcuticular Surgical Suture (N=171) | Surgical Staples (N=179)
infection at 4 - 6 weeks post delivery (Infections and infestations) | 6 | 4
disruption of wound at 4 - 6 weeks post delivery (Skin and subcutaneous tissue disorders) | 6 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No